CLINICAL TRIAL: NCT03885999
Title: Functional Anorectal Studies in Patients With Low Anterior Resection Syndrome (LARS)
Brief Title: Studies in Patients With Low Anterior Resection Syndrome (LARS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giome (Other)
Responsible Party: Principal Investigator, Hans Gregersen, Professor, Giome
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018.640
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Anterior Resection Syndrome; Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecobionics studies (Experimental)
  Interventions: Device: Fecobionics

INTERVENTIONS:
Device: Fecobionics — Fecobionics is a new device for studying defecation

SUMMARY:
Colorectal Cancer is the commonest cancer diagnosed for both genders combined in Hong Kong. In 2015 16.6% of all new cancer cases registered on the Hong Kong registry were cancer of colon and rectum. With recent development in oncological and surgical treatments for rectal cancer, many patients are receiving sphincter-preserving surgery with low colorectal or coloanal anastomosis to avoid permanent stoma.

Up to 80% of patients who has undergone low anterior resection (LAR), suffer from severe bowel dysfunction post operatively. Patients may suffer from a wide range of symptoms from incontinence, frequency, and urgency to constipation and feelings of incomplete emptying. This combination of symptoms after LAR is referred to as Low Anterior Resection Syndrome (LARS) which is associated with negative impact on quality of life (QoL). Originally, it was thought that these symptoms were due to early postoperative changes. Many studies report that the majority of patients experience longterm changes in quality of life after LAR. Therefore, a large number of patients worldwide are suffering from unpredictable, poor bowel function postoperatively affecting their day-to-day activity and quality of life. The cause of LARS is often multifactorial and difficult to define. Unfortunately, there is no cure for LARS at present. This trial is designed to use Fecobionics, a new Hong Kong based innovation of a simulated stool, to provide new mechanistic insights regarding anorectal physiological function post low anterior resection to understand the condition better to improve their treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with history of LARS over 3 months.
* Informed, written consent by the patient

Exclusion Criteria:

* Patients who are not willing to undergo the specified tests in this study
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at at Prince of Wales Hospital in Hong Kong from 29 May 2019 to 9 December 2019. The protocol was approved by the Ethics Review Committees of the involved hospital (CRE-2018.640). Written informed consent was obtained from each subject prior to commencement of the study.
Period: Overall Study
Arm/Group | Fecobionics Studies
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fecobionics Studies
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Patients attending the colorectal functional clinic Prince of Wales Hospital in Hong Kong for management of severe low anterior resection syndrome post anterior resection for treatment of rectal cancer were invited to join this exploratory study.
  Participants
    Hong Kong | 11
LARS score [Median (Inter-Quartile Range); unit: units on a scale] — The Low anterior resection syndrome score system was based on the published paper(Katrine J Emmertsen & Laurberg, 2012). The range of the score (0-42) was divided into groups of 0 to 20 (no LARS), 21 to 29 (minor LARS), and 30 to 42 (major LARS).
  units on a scale | 39 [38.5 to 39.5]

OUTCOME MEASURES:

1. Primary Outcome: Change of Anorectal Pressure Assessed With the Fecobionics Device
Description: The expected outcome is that the device will perform as shown in the previous human experiments (n>60) where no adverse effects have been recorded.
Time Frame: baseline and following intervention, approximately 30 seconds
Population: 11 LARS patients
Measure: Mean (Standard Error); unit: cmH2O
Arm/Group | Fecobionics Studies
Number analyzed (Participants) | 11
cmH2O | 9.8 (2.1)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Same definitions as the clinicaltrials.gov.
Arm/Group | Fecobionics Studies
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fecobionics Studies (N=12)
Perforation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03885999/Prot_SAP_000.pdf